CLINICAL TRIAL: NCT07333586
Title: Insomnia, Metabolic Syndrome and Insulin Resistance
Brief Title: Insomnia and Insulin Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: insomnia
Record Dates: First submitted 2025-12-02; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Insulin Resistance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-1 (Active Comparator): treatment with cognitive behavior therapy for insomnia this is behaviorial therapy that meets with a "coach" once a week for 5 wk
  Interventions: Behavioral: CBT-I
- sleep hygiene (Placebo Comparator): treatment with sleep hygiene group meets with a coach once at the beginning of the intervention period
  Interventions: Behavioral: sleep hygiene

INTERVENTIONS:
Behavioral: CBT-I — meets with "coach" who is teaching the participant how to deal with insomnia meets 5 times/once a week with the coach
  Arms: CBT-1
Behavioral: sleep hygiene — meets with coach 1 time and is teaching the participant how to improve their sleep
  Arms: sleep hygiene

SUMMARY:
Insomnia symptoms are linked to metabolic syndrome (MetS), which includes abnormal glucose metabolism, insulin resistance (IR), and incidence of diabetes. Chronic sleep deficit is a major predictor of disease and early mortality. Further, insomnia is the most common sleep disorder in the United States. The recommended first line of treatment for insomnia is Cognitive Behavioral Therapy for Insomnia (CBT-I). CBT-I is a multidimensional treatment that targets the thoughts and behaviors that perpetuate insomnia symptoms over time. This study will explore CBT-I effects on MetS outcomes (ie. blood pressure, triglycerides, etc.) and provide preliminary evidence that CBT-I impacts IR and fasting glucose concentrations within this population.

20 subjects with insomnia will be recruited. They will be randomly assigned to either CBT-i or sleep hygiene. The intervention is 5 wks. Pre and post intervention, the investigator will have participants fill out a number of questionnaires, a daily sleep diary, 2 weeks of actigraphy measuring sleep and physical activity and there will be a single blood draw at the beginning and the end of the study.

DETAILED DESCRIPTION:
Insomnia symptoms are linked to metabolic syndrome (MetS), which includes abnormal glucose metabolism, insulin resistance (IR), and incidence of diabetes. In young healthy individuals, shortened sleep duration results in IR and elevated free fatty acid concentrations and has been associated with circadian misalignment. Additionally, individuals with type 2 diabetes (T2D) frequently have insufficient sleep or poor sleep quality, and greater sleep disturbances are associated with poorer glycemic control. Thus chronic sleep deficit is a major predictor of disease and early mortality. Further, insomnia is the most common sleep disorder in the United States, impacting at least 10% of the general population and ~40% of those with T2D. Although stress or changes in lifestyle habits often cause short-term insomnia, chronic insomnia (Insomnia Disorder) is defined as difficulty falling or staying asleep that causes daytime impairment 3 or more nights a week, lasts 3 or more months, and cannot be fully explained by another health problem.

The recommended first line of treatment for insomnia is Cognitive Behavioral Therapy for Insomnia (CBT-I). CBT-I is a multidimensional treatment that targets the thoughts and behaviors that perpetuate insomnia symptoms over time. The cognitive components of the therapy empower patients to challenge their automatic thoughts and reactions to poor sleep, and the behavioral components focus on matching time in bed to sleep ability in order to increase homeostatic sleep drive (or natural propensity for sleep). CBT-I improves insomnia in many populations (e.g., among those with psychological and physical comorbidities, chronic pain, etc). CBT-I has also demonstrated efficacy in reducing insomnia symptoms among those with IR in two pilot studies, but no studies have been powered to test CBT-I effects on metabolic outcomes within this population.

Obesity is a leading risk factor for impaired metabolic health. Given the impact of insomnia symptoms on MetS, effective treatment of insomnia may improve metabolic outcomes among those with obesity. This study aims to:

1. Demonstrate the feasibility of the proposed CBT-I protocol. Specifically, the investigators hypothesize that ≥85% of participants will complete all assigned treatment sessions and follow-ups.
2. Replicate previous findings that CBT-I reduces insomnia among obese adults with insomnia.
3. Explore CBT-I effects on MetS outcomes (ie. blood pressure, triglycerides, etc.).
4. Provide preliminary evidence that CBT-I impacts IR and fasting glucose concentrations within this population.

20 subjects with insomnia will be recruited. Participants will be randomly assigned to either CBT-i or sleep hygiene. The intervention is 5 wks. Pre and post intervention, the investigators will have participants fill out a number of questionnaires, a daily sleep diary, 2 weeks of actigraphy measuring sleep and physical activity and there will be a single blood draw at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

ages 18-50 y BMI 28-45 kg/m2 Score on the Insomnia Severity Index ≥15.

Exclusion Criteria:

contraindications for CBT-I (mania or seizure disorder) symptoms requiring immediate attention (e.g., psychosis, suicide intent) report illicit substance use on a monthly basis (e.g., cocaine, opioids) receiving behavioral treatment for insomnia overt cardiovascular disease overt renal disease thyroid disease cancer pregnant dieting using GLP-1 agonists taking exogenous insulin

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
insulin resistance | baseline and through study completion, an average of 9 weeks
  HOMA-IR calculation

SECONDARY OUTCOMES:
sleep duration | baseline and through study completion, an average of 9 weeks
  measuring sleep duration with Actigraph

IPD SHARING:
Plan to Share IPD: Yes